CLINICAL TRIAL: NCT05343312
Title: Monitoring the Therapeutic Efficacy of the Combinations Artemether-Lumefantrine, Amodiaquine-Artesunate, Dihydroartemisinin-Piperaquine, and Pironaridine-Artesunate in the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Children Under 5 Years of Age in Five Sentinel Sites in Mozambique
Brief Title: In Vivo Efficacy of Artemether-Lumefantrine, Amodiaquine-Artesunate, Dihydroartemisinin-Piperaquine, and Pironaridine-Artesunate in Mozambique
Acronym: MEFI_IV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de Investigacao em Saude de Manhica (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/CNBS/22
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Malaria
Keywords: Treatment; Artemisine-based combinations; children
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Artemether-Lumefantrine (AL) (Active Comparator): AL (Coartem™) will be administered twice daily for three days (six doses in total) with dosage determined according to body weight: one tablet (20mg artemether and 120mg lumefantrine) for children 5 to <15kg, two tablets per dose for those 15 to <25kg, and three tablets per dose for those 25 to <35kg.
  Interventions: Drug: AL (Coartem)
- Amodiaquine-Artesunate (AS-AQ) (Active Comparator): AQ-AS (Coarsucam™) will be administered once daily according to body weight: one 25mg artesunate and 67.5mg amodiaquine tablet in children <9kg, one 50mg artesunate and 135mg amodiaquine tablet in children 9-17.9kg; and one 100mg artesunate and 270mg amodiaquine tablet in children >18-35kg.
  Interventions: Drug: AS-AQ (Carsucam)
- Dihydroartimisin+Piperaquine (DHP) (Active Comparator): DHP will be administered once daily according to body weight: tablet (40 mg dihydroartimisin+artesunate) half in children 5 < 10kg, one in children 10 < 20kg and 2 tablets for those children over 20 kg.
  Interventions: Drug: DHP
- Pyronaridine +Artesunate (PA) (Active Comparator): PA will be administered once daily according to body weight: granule ( 60 mg pyronaridine + 20 artesunate), one in children 5 < 7kg, two in children 8 < 15kg and three in children 15 < 20kg. Tablets ( 180 mg pyronaridine+ 60 mg artesunate), one in children 20 < 24Kg and two in children 24 < 45Kg.
  Interventions: Drug: PA

INTERVENTIONS:
Drug: AL (Coartem) — Eligible patients will be consecutively assigned to the four cohorts. Rescue therapy according to national malaria treatment guidelines will be also administered in cases of early or late treatment failure.
  Follow-up visits will take place on days 1, 2, 3, 7, 14,21 and 28 after enrolment or at any time point whenever the child is sick. Adverse events will be recorded and assessed for severity and association with study medication.
  Thick and thin Giemsa-stained blood slides will be prepared before each dose to be administered and at every follow-up visit of days 2, 3, 7, 14, 21, 28, 35 and 42. Blood samples for PCR analysis will be collected from every patient at baseline and at days 7, 14, 28, and 42 day of treatment failure or at any other unscheduled visit. The Molecular markers associated with suboptimal response to ACTs will be investigated.
  Arms: Artemether-Lumefantrine (AL)
Drug: AS-AQ (Carsucam) — Eligible patients will be consecutively assigned to the four cohorts. Rescue therapy according to national malaria treatment guidelines will be also administered in cases of early or late treatment failure.
  Follow-up visits will take place on days 1, 2, 3, 7, 14,21, 28, 35 and 42 after enrolment or at any time point whenever the child is sick. Adverse events will be recorded and assessed for severity and association with study medication.
  Thick and thin Giemsa-stained blood slides will be prepared before each dose to be administered and at every follow-up visit of days 2, 3, 7, 14, 21, 28, 35 and 42. Blood samples for PCR analysis will be collected from every patient at baseline and at days 7, 14, and 28 day of treatment failure or at any other unscheduled visit. The Molecular markers associated with suboptimal response to ACTs will be investigated.
  Arms: Amodiaquine-Artesunate (AS-AQ)
Drug: DHP — Eligible patients will be consecutively assigned to the four cohorts. Rescue therapy according to national malaria treatment guidelines will be also administered in cases of early or late treatment failure.
  Follow-up visits will take place on days 1, 2, 3, 7, 14,21, 28, 35 and 42 after enrolment or at any time point whenever the child is sick. Adverse events will be recorded and assessed for severity and association with study medication.
  Thick and thin Giemsa-stained blood slides will be prepared before each dose to be administered and at every follow-up visit of days 2, 3, 7, 14, 21, 28, 35 and 42. Blood samples for PCR analysis will be collected from every patient at baseline and at days 7, 14, 28, and 42 day of treatment failure or at any other unscheduled visit. The Molecular markers associated with suboptimal response to ACTs will be investigated.
  Arms: Dihydroartimisin+Piperaquine (DHP)
Drug: PA — Eligible patients will be consecutively assigned to the four cohorts. Rescue therapy according to national malaria treatment guidelines will be also administered in cases of early or late treatment failure.
  Follow-up visits will take place on days 1, 2, 3, 7, 14,21, 28, 35 and 42 after enrolment or at any time point whenever the child is sick. Adverse events will be recorded and assessed for severity and association with study medication.
  Thick and thin Giemsa-stained blood slides will be prepared before each dose to be administered and at every follow-up visit of days 2, 3, 7, 14, 21, 28, 35 and 42. Blood samples for PCR analysis will be collected from every patient at baseline and at days 7, 14, 28, and 42 day of treatment failure or at any other unscheduled visit. The Molecular markers associated with suboptimal response to ACTs will be investigated.
  Arms: Pyronaridine +Artesunate (PA)

SUMMARY:
This is a classical in vivo clinical trial, following World Health organization's recommendations, ran as a multisite study within Mozambique trying to assess the efficacy and safety in 5 sites of the four oral ACTS artemether-lumefantrine (AL), Amodiaquine-Artesunate (AQ-AS), Dihydroartemisinin-Piperaquine (DHP) and Pironaridine-Artesunate for the treatment of uncomplicated malaria in children aged<5 years.

DETAILED DESCRIPTION:
Eligible patients were consecutively assigned to the cohort and treated with AL (cohort 1), AQ-AS (cohort 2), DHP (cohort 3) and PA (cohort 4). AL (Coartem™) will be administered twice daily for three days (six doses in total) with dosage determined according to body weight: one tablet (20mg artemether and 120mg lumefantrine) for children 5 to <15kg, two tablets per dose for those 15 to <25kg, and three tablets per dose for those 25 to <35kg. AQ-AS (Winthrop™) will be administered once daily according to body weight: one 25mg artesunate and 67.5mg amodiaquine tablet in children <9kg, one 50mg artesunate and 135mg amodiaquine tablet in children 9-17.9kg; and one 100mg artesunate and 270mg amodiaquine tablet in children >18-35kg. DHP will be administered once daily according to body weight: half tablet (40mg dihydroartemisinin e 320 mg piperaquine) for children 5 to < 10Kg, one tablet for per dose for those 10 < 20Kg and 2 tablets for 20 or more Kg. PA (granules 60mg pirinaridine +/20mg artesunate) will administered once daily according to body weight: 1 granule per dose for children 5 to < 8Kg, two for children 8 < 15Kg, three for those 15 < 20Kg. PA (180mg pyrinaridine+60 mg artesunate) one tablet for children 20 < 24Kg and two tablets for those 24 < 45Kg. All treatments will be directly observed for a minimum of 30 minutes. Vomiting occurring within the first 30 minutes implied the repetition of the full dose of treatment. For those patients living far away from the health facilities, and for which direct observation of the evening doses of AL was challenging, admission was offered for the first three days of the study.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6 to 59 months
* Weight Greater than or equal to 5 kg
* Absence of severe malnutrition;
* Mono-infection with Plasmodium falciparum in blood, confirmed by microscopy;
* Parasite density between 2,000 and 200,000 asexual parasites per microliter of blood;
* Axillary temperature ≥ 37.5 C° or history of fever in the last 24 hours;
* Lack of danger signs, or no signs of severe and / or complicated malaria according to the WHO definition
* Ability to swallow the drugs
* Haemoglobin greater than 5.0 g / dl
* Residents within the study area and have the possibility of an adequate follow-up in the days of monitoring for a period of 28 days;
* Absence of a history of hypersensitivity to study medications;
* Informed consent of parents, guardians or caregivers (legal guardian) after explaining the purpose of the study.

Exclusion Criteria:

* Presence of any danger sign or severe or complicated Plasmodium falciparum malaria according to WHO definitions
* Presence of fever due to diseases other than malaria (eg measles, acute respiratory infection, severe diarrhea with dehydration) or other known diseases, with chronic or serious illnesses (cardiac, renal, hepatic or known infection with HIV AIDS),
* Presence of severe malnutrition (defined as a child whose growth pattern is below the 3rd percentile, mid-upper-arm circumference <110mm, weight / height <70% according to the WHO tables, or the presence of bilateral edema of the lower limbs)
* Multi or mono-infection by another Plasmodium species detected by microscopy;
* Regular medication that may interfere with the pharmacokinetics of antimalarials;
* History of hypersensitivity or contraindication to study drug;
* A history of taking antimalarial drugs or drugs with antimalarial activity in less than 7 days.
* Continuous prophylaxis with cotrimoxazole in HIV positive children

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 870 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
To measure the Day 28, PCR corrected cure rates of artemether-lumefantrine and Amodiaquine-artesunate. | 28 days
  This cure rate is defined as the proportion of patients with adequate clinical and parasitological response (ACPR) at Day 28, once PCR correction to differentiate recrudescences from new infections have been applied (and hence only considering as treatment failures those parasite recurrences confirmed as recrudescences).
To measure the Day 42, PCR corrected cure rates of Dihydroartemisinin-Piperaquine and Pironaridine-Artesunate | 42 days
  This cure rate is defined as the proportion of patients with adequate clinical and parasitological response (ACPR) at Day 42, once PCR correction to differentiate recrudescences from new infections have been applied (and hence only considering as treatment failures those parasite recurrences confirmed as recrudescences).

SECONDARY OUTCOMES:
To evaluate the incidence of adverse events | 28/42 days
  Safety was assessed by administering a questionnaire about the nature and incidence of adverse events and serious adverse events. An adverse event is defined as any unfavorable, unintended sign, symptom, syndrome or disease that develops or worsens with the use of a medicinal product, regardless of whether it is related to the medicinal product.
To measure the Day PCR uncorrected cure rates of Artemether-Lumefantrine, Amodiaquine-Artesunate, Dihydroartemisinin-Piperaquine, and Pironaridine-Artesunate. | 28/42 days
  This cure rate is defined as the proportion of patients with adequate clinical and parasitological response (ACPR) at Day 28/42, without PCR correction to differentiate recrudescences from new infections and hence considering as treatment failures all parasite recurrences.
Evaluate the presence of Molecular Markers associated with sub optimum responses to ACTs | 28/42 days
  The presence of molecular marks is defined as presence of mutations in pfk13 and pfmdr1 (at codons 86, 184 and 1246) genes identified by Sanger sequencing of pre-treatment samples.

CONTACTS AND LOCATIONS:
Locations (5):
- Mozambique (5):
  - Hospital Rural de Montepuez, Montepuez, Cabo Delgado Province
  - Hospital Distrital de Mssinga, Massinga, Inhambane Province
  - Hospital Distrital de Dondo, Dondo, Sofala
  - Mospital Distrital de Moatize, Moatize, Tete
  - Hospital Distrital de Mopeia, Mopeia, Zambezia Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nhama A, Chidimatembue A, Nhamussua L, Bassat Q, da Silva C, Nhacolo A, Arnaldo P, Salvador C, Cassy A, Candrinho B, Dimene M, Carvalho E, Saifodine A, Wate F, Mucavele H, Torres-Mendoza Y, Horton B, Plucinski M, Cistero P, Mayor A, Aide P. Efficacy of artemether-lumefantrine, artesunate-amodiaquine, dihydroartemisinin-piperaquine and artesunate-pyronaridine for the treatment of uncomplicated Plasmodium falciparum malaria in Mozambique, 2022. Malar J. 2025 Jul 14;24(1):231. doi: 10.1186/s12936-025-05473-9. PMID 40660279
- See also: Related Info — http://www.cismmanhica.org